CLINICAL TRIAL: NCT01425606
Title: a Study to Evaluate the Electrolyte Changes in Particular Sodium,in Multiple Myeloma and the Effect of the m- Proteins on the Strong Ion Difference
Brief Title: Pseudohyponatremia of Multiple Myeloma is True Hyponatremia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 039-2011
Record Dates: First submitted 2011-06-09; First posted 2011-08-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Hyponatremia of Multiple Myeloma
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- blood test: to measure levels of sodium, albumin and acid - base status in venous blood
  Interventions: Other: blood test

INTERVENTIONS:
Other: blood test — blood test to measure levels of: sodium, albumin and acid - base status in venous blood.

SUMMARY:
Hypothesis: the hyponatremia of multiple myeloma (m.m.)is true and not pseudohyponatremia by using the stewart approach to acid - base interpretation, would like to show that the positive charged m- proteins produced in m.m.result in true hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* patients with multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with gammaglobulinemia and\or multiple myeloma.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
hyponatremia present or not | one year
hyponatremia | one year
  pseoudohyponatremia or not

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Hospital, Kfar Saba, Israel